CLINICAL TRIAL: NCT02282696
Title: Research on Psychosocial Aspects in the Care for Patients With Cancer: Validation Study CARES.
Brief Title: Validation Study CARES
Acronym: OPSA-PK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Vrije Universiteit Brussel (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Johan Hellings, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPSA-PK
Record Dates: First submitted 2014-07-16; First posted 2014-11-04 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cancer patients (Experimental): Questionnaire, focus group participation
  Interventions: Other: Questionnaire, focus group participation

INTERVENTIONS:
Other: Questionnaire, focus group participation — participants of the quantitative part of the study are asked to fill in a questionnaire, participants of the qualitative part are asked to participate in a focus group interview.

SUMMARY:
This study aims to validate the CARES, a needs assessment instrument which can be used to inventorize cancer patients biopsychosocial distress and care needs.

* QUANTITATIVE PART OF THE STUDY: Patients need to fill in a questionnaire package containing questions about social-demographic and medical data, the CARES and convergent measures: Karnofsky Performance Scale (KPS), Hospital Anxiety Depression Scale (HADS), Social Support List (SSL), Maudsley Marital Questionnaire (MMQ), European Organisation for Research and Treatment of Cancer Quality Of Life Core 30 (EORTC-QOL-C30), Distress Thermometer (DT) and a Care Needs Questionnaire. One week after the first questionnaire package participants have to fill in the CARES a second time and answer some questions to evaluate the feasibility of the CARES.
* QUALITATIVE PART OF THE STUDY: Participants from the quantitative part of the study and other (ex-) cancer patients who not have to fulfill the criteria of age and cancer stage can participate in a focus group interview. In these focus groups the content validity and preferences on psychosocial screening in care are discussed.

ELIGIBILITY:
Inclusion Criteria:

* Primary cancer diagnosis stage I, II, III
* All types of cancer

Exclusion Criteria:

* Having had or premorbid neurological problems or cognitive dysfunctions.
* The lack of proficiency in Dutch (Flemish).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Validity of the CARES | week 1
  CARES-total and subscale scores. Computation of internal consistency of summary scales (for reliability), intra-class correlation between test and retest scores (for reliability), confirmatory factor analysis (for construct-validity)
Convergent validity of the CARES | week 1
  Total- and subscale scores of convergent instruments (KPS, HADS,SSL, MMQ, EORTC-QOL-C30, DT). Computation of correlation between CARES-scores and scores of convergent instruments.

SECONDARY OUTCOMES:
To assess the distress and care needs of cancer patients | week 1
  inventorization of level of distress, number and kind of difficulties and care needs experienced by cancer patients
To assess patients experiences with psychosocial care | week 1
  Patients experiences of the approach of psychosocial wellbeing in cancer care, and their preferences in this area.

CONTACTS AND LOCATIONS:
Overall Officials: Hellings Johan, Principal Investigator — Hasselt University; Bojoura Schouten, dra., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

REFERENCES:
- [Derived] Schouten B, Hellings J, Van Hoof E, Vankrunkelsven P, Bulens P, Buntinx F, Mebis J, Vandijck D, Schrooten W. Validation of the flemish CARES, a quality of life and needs assessment tool for cancer care. BMC Cancer. 2016 Aug 30;16(1):696. doi: 10.1186/s12885-016-2728-9. PMID 27576341
- [Derived] Schouten B, Van Hoof E, Vankrunkelsven P, Schrooten W, Bulens P, Buntinx F, Mebis J, Vandijck D, Cleemput I, Hellings J. Assessing cancer patients' quality of life and supportive care needs: Translation-revalidation of the CARES in Flemish and exhaustive evaluation of concurrent validity. BMC Health Serv Res. 2016 Mar 11;16:86. doi: 10.1186/s12913-016-1335-4. PMID 26969509